CLINICAL TRIAL: NCT02576678
Title: A Phase 2, Multicenter, Open-Label Study to Assess the Safety, Tolerability and Pharmacokinetics of Apremilast (CC-10004) in Pediatric Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study of Safety, Tolerability and Pharmacokinetics of Apremilast (CC-10004) in Pediatric Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-10004-PPSO-001
Expanded Access: NCT03740516 (No longer available)
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Psoriasis
Keywords: Psoriasis; Moderate to Severe Plaque Psoriasis; Plaque Psoriasis; CC-10004; Apremilast; Pharmacokinetics; Open-label; Safety; Pediatric
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open label apremilast (Experimental): Apremilast doses of 10-mg, 20-mg or 30-mg tablets have been selected to determine the dose range in adolescents and children with moderate to severe plaque psoriasis. These pediatric dosages are expected to achieve exposures similar to those achieved in adult psoriasis and psoriatic arthritis (PsA) subjects treated with apremilast 30 mg orally twice daily (BID).
  A staggered, stepwise approach by age range and weight (starting with older and heavier subjects) is considered appropriate for this first-time-in-children study. Doses for younger and lower body weight subjects will be adjusted based on safety and PK data from older and heavier subjects.
  Subjects will be divided into 2 age groups with at least 16 subjects in each group. Dosing within and between groups will be staggered, based on PK data collected and on a minimum of 2 weeks of safety data.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast
  Other Names: CC-10004

SUMMARY:
This is a Phase 2, multicenter, open-label study in subjects with moderate to severe plaque psoriasis aged 6 to 17 years, inclusive, intended to assess the safety, tolerability, and PK of apremilast with 2 weeks of oral apremilast treatment followed by a 48-week extension of apremilast treatment. Moderate to severe plaque psoriasis is defined as Psoriasis Area Severity Index (PASI) ≥ 12, Body Surface Area (BSA) ≥ 10%, and static Physician Global Assessment (sPGA) of ≥ 3. The total study duration for each subject will last for up to a total of 107 weeks which includes screening, treatment (including the PK portion of the study and the extension treatment period), two short-term follow-up periods and a long-term follow-up period.

DETAILED DESCRIPTION:
Each subject will undergo a screening period of up to 5 weeks, a treatment period of 2 weeks with PK sample collection, and an extension treatment period of 48 weeks, to allow subjects access to apremilast treatment if medically appropriate (following the completion of the 2 week PK portion). Regardless of when they stop treatment, subjects should complete two post treatment follow-up visits at approximately 4 and 8 weeks after the last dose. All subjects should complete the final follow-up visit at Week 102 or at a timepoint 52 weeks after the last dose of apremilast was taken in subjects who have withdrawn at any time prior to Week 50. At least 32 subjects will be enrolled into this study to provide an adequate PK profile and safety assessment in subjects of different ages and body weight ranges. Subjects will be divided into 2 age groups (adolescents [ages 12 to 17 years, inclusive] and children [ages 6 to 11 years, inclusive]), with at least 16 subjects in each group. Apremilast treatment will start in older and heavier subjects.

Group 1 (ages 12 to 17 years, inclusive; weight ≥ 35 kg)

* The data collected from the first 8 subjects will be reviewed by an independent data monitoring committee (DMC) to determine if it is appropriate to proceed with dosing the balance of Group 1 subjects and to proceed with dosing in the Group 2 subjects.

and an evaluation of these data by the DMC has been completed.

Group 2 (ages 6 to 11 years, inclusive; weight ≥ 15 kg)

* The dose regimens (dose strength and/or dose frequency) for these first 8 subjects will be based upon the PK and safety assessments from the first 8 subjects in Group 1.
* For the remaining subjects in Group 2, the dose (dose strength and/or dose frequency) will be based upon the subject weight as determined by the PK and safety assessments. The dose strength and/or dose frequency will be adjusted for any safety concerns or for unexpected changes in exposure. In the event of a dose regimen adjustment after the second PK and safety assessment, the first 8 subjects in Group 2 will return to the site for the appropriate dosing adjustment.

ELIGIBILITY:
Inclusion Criteria:

- Subjects must satisfy all of the following criteria to be enrolled in the study:

1. Male or female subjects 6 to 17 years of age, inclusive, at the time the informed consent document is signed by the legal guardian
2. Group 1 Only: ages 12 to 17 years, inclusive, and weighs ≥ 35 kg
3. Group 2 Only: ages 6 to 11 years, inclusive, and weighs ≥ 15 kg
4. Subject is able to swallow the apremilast tablet
5. Able to sign an assent with a legal guardian who can understand and voluntarily sign an informed consent
6. Able to adhere to the study visit schedule and other protocol requirements
7. Must agree to withhold vaccinations during the first 2 weeks of dosing. Inactivated vaccines will be allowed during the extension treatment period
8. Diagnosis of chronic plaque psoriasis for at least 6 months prior to Screening
9. Have moderate to severe plaque psoriasis at Screening and Baseline as defined by:

   * Psoriasis Area and Severity Index (PASI) score ≥ 12; and
   * Body surface area (BSA) ≥ 10%; and
   * Static Physician Global Assessment (sPGA) ≥ 3 (moderate to severe)
10. Disease inadequately controlled by or inappropriate for topical therapy for psoriasis
11. Candidate for systemic or phototherapy
12. Have not been exposed to any or have been exposed to no more than one systemic agent for psoriasis
13. At Screening, laboratory values must be within the following ranges:

    * White blood cell (WBC) count Age (yrs) Males (x 103 /µL) Females (x 103 /µL) 6-11 3.5 - 13.65 3.5 - 13.65 12-18 3.5 - 13.15 3.5 - 13.15
    * Platelet count Age (yrs) Males (x 103 /µL) Females (x 103 /µL) 6-11 117 - 394 117 - 394 12-18 126 - 400 126 - 400
    * Hemoglobin (Hb) Age (yrs) Males (g/dL) Females (g/dL) 6-11 10.0 - 15.5 10.0 - 15.5 12-18 11.0 - 18.1 10.0 - 16.4
14. Male subjects who engage in activity in which conception is possible must use barrier contraception (male latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]) while on apremilast and for at least 28 days after the last dose of apremilast
15. All females of childbearing potential (FCBP) must either practice abstinence* from heterosexual contact or use one of the approved contraceptive options as described below while on apremilast and for at least 28 days after dministration of the last dose of apremilast. For the purposes of this study, a female subject is considered of childbearing potential if she is ≥ 12 years old or has reached menarche, whichever occurred first At the time of study entry, and at any time during the study when a female subject of childbearing potential's contraceptive measures or ability to become pregnant changes, the Investigator will educate the subject regarding abstinence or contraception options and the correct and consistent use of effective contraceptive methods in order to successfully prevent pregnancy Females of childbearing potential must have a negative pregnancy test at Screening and Baseline. All FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below: Option 1: Any one of the following effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide * Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* The presence of any of the following will exclude a subject from enrollment:

  1. History of or currently active inflammatory bowel disease
  2. Major concurrent medical conditions, pregnancy or lactation
  3. Any condition that confounds the ability to interpret data from the study
  4. Guttate, erythrodermic, or pustular psoriasis
  5. Psoriasis flare or rebound within 4 weeks prior to Screening
  6. Evidence of skin conditions that would interfere with clinical assessments
  7. History of human immunodeficiency virus infection, or positive result to hepatitis B surface antigen or hepatitis C antibodies at Screening
  8. Clinically significant abnormality on 12-Lead ECG at Screening
  9. History of active mycobacterial infection with any species (including Mycobacterium tuberculosis) within 3 years of the Screening Visit and without documentation of successful treatment
  10. Congenital and acquired immunodeficiencies (eg, Common Variable Immunodeficiency),immunoglobulin A deficiency
  11. History of recurrent significant infections
  12. Active infection or infection treated with antibiotic treatment within 2 weeks of first dose
  13. Any history of or active malignancy
  14. History of allergy/intolerance to any component of the investigational product, ie, apremilast, lactose monohydrate, microcrystalline cellulose, croscarmellose sodium, magnesium stearate, hypromellose 15 cP, titanium dioxide, polydextrose FCC, talc, maltodextrin, medium chain triglycerides, iron oxide red, iron oxide yellow, and iron oxide black.
  15. Deficiencies in lactose metabolism, ie, galactose-1-phosphate uridylyltransferase, UDPglactose 4-epimerase, galactokinase or Fanconi Bickel syndrome, including congenital lactase deficiencies, and glucose-galactose malabsorption.
  16. Any other significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study or which places the subject at unacceptable risk if he/she were to participate in the study
  17. Prior history of suicide attempt at any time in the subject's lifetime prior to screening or enrollment in the study or major psychiatric illness requiring hospitalization within 3 years
  18. Answering '"Yes'" to any question on the Columbia-Suicide Severity Rating Scale during screening or at baseline
  19. Having received biologic therapy within 5 terminal half-lives, including but not limited to the following time periods:

      * Four weeks prior to baseline for etanercept
      * Ten weeks prior to baseline for adalimumab
      * Twenty-four weeks prior to baseline for ustekinumab
  20. Topical therapy within 2 weeks of baseline (including but not limited to topical corticosteroids, topical retinoid or vitamin D analog preparations, tacrolimus, pimecrolimus, or anthralin/dithranol)

      * Exceptions: low-potency corticosteroids (please refer to the Investigators' Manual) will be allowed as background therapy for treatment of the face, axillae, and groin in accordance with the manufacturers' suggested usage during the course of the study
      * Subjects with scalp psoriasis will be permitted to use coal tar shampoo and/or salicylic acid scalp preparations on scalp lesions
      * An unmedicated skin moisturizer (eg, Eucerin®) will be also permitted for body lesions only. Subjects should not use these topical treatments within 24 hours prior to the clinic visit
  21. Systemic therapy for psoriasis within 4 weeks prior to baseline (including but not limited to cyclosporine, corticosteroids, methotrexate, oral retinoids, mycophenolate, thioguanine, hydroxyurea, sirolimus, sulfasalazine, azathioprine, and fumaric acid esters)
  22. Use of phototherapy (ie, UVB, PUVA)within 4 weeks prior to baseline
  23. Use of any investigational drug within 4 weeks prior to baseline, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer)
  24. Children in Care: a child who has been placed under the control or protection of an agency, organization, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation
  25. Prior treatment with apremilast

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2019-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (18):
- United States (6):
  - Rady Children's Hospital, San Diego, California
  - Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago Department of Dermatology, Chicago, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - Mount Sinai, St. Luke's, New York, New York
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
- Canada (3):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - CHU Saint-Justine, Montreal, Quebec
- Germany (6):
  - Rheinische Friedrich-Wilhelms-Universitaet Bonn - Universitaetsklinikum Bonn, Bonn
  - Universitatsklinikum Essen, Essen
  - Universitatsklinikum Klinikum Frankfurt Main, Frankfurt
  - Kinderkrankenhaus Wilhelmstift, Dermatologie, Hamburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Muenster University Hospital (Universitätsklinikum Muenster), Münster
- Spain (3):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Sant Joan de Deu, Esplugues de Llobregat
  - Hospital La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Result] Paller AS, Hong Y, Becker EM, de Lucas R, Paris M, Zhang W, Zhang Z, Barcellona C, Maes P, Fiorillo L. Pharmacokinetics and safety of apremilast in pediatric patients with moderate to severe plaque psoriasis: Results from a phase 2 open-label study. J Am Acad Dermatol. 2020 Feb;82(2):389-397. doi: 10.1016/j.jaad.2019.08.019. Epub 2019 Aug 10. PMID 31408686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 11 study centers in 4 countries, including the United States, Canada, Germany and Spain.
Pre-assignment Details: Participants were enrolled according to a staggered, stepwise approach by age range and weight starting with older and heavier participants. Dosing within and between groups was staggered based on PK data collected and a minimum of 2 weeks of safety data.
Groups:
- Group 1 Adolescents: Apremilast 20 mg: Participants ages 12 to 17 years old, with a weight of ≥ 35 kg to < 70 kg received apremilast tablets 20 mg twice a day (BID) for 2 weeks followed by a 48-week extension of apremilast treatment.
- Group 1 Adolescents: Apremilast 30 mg: Participants ages 12 to 17 years old, with a weight of ≥ 70 kg received apremilast 30 mg tablets BID for 2 weeks followed by a 48-week extension of apremilast treatment.
- Group 2 Children: Apremilast 20 mg: Participants ages 6 to 11 years old, with a weight of ≥ 15 kg received apremilast 20 mg tablets BID for 2 weeks followed by a 48-week extension of apremilast treatment.
Period: Overall Study
Arm/Group | Group 1 Adolescents: Apremilast 20 mg | Group 1 Adolescents: Apremilast 30 mg | Group 2 Children: Apremilast 20 mg
Started | 13 | 8 | 21
Pharmacokinetic (PK) Population (PK participants had at least 1 dose of drug and had evaluable PK data) | 12 | 8 | 18
Completed (Completed = participants who completed week 50.) | 8 | 7 | 16
Not Completed | 5 | 1 | 5
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Withdrawal by Subject | 3 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Miscellaneous | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population consisted of all participants who were enrolled and received at least 1 dose of apremilast.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Adolescents: Apremilast 20 mg | Group 1 Adolescents: Apremilast 30 mg | Group 2 Children: Apremilast 20 mg | Total
Number analyzed (Participants) | 13 | 8 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.8 (1.77) | 14.8 (2.05) | 9.3 (1.35) | 11.8 (2.95)
Age, Customized [Count of Participants; unit: Participants]
  6 to 11 years | 0 | 0 | 21 | 21
  12 to 17 years | 13 | 8 | 0 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 13 | 23
  Male | 4 | 7 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 5 | 9
  Not Hispanic or Latino | 12 | 5 | 16 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 2 | 4
  Black or African American | 0 | 0 | 2 | 2
  Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 1
  White or Caucasian | 10 | 6 | 16 | 32
  Other | 1 | 1 | 1 | 3
Baseline Weight Category (kg) [Count of Participants; unit: Participants]
  < 15 kg | 0 | 0 | 0 | 0
  ≥ 15 - < 35 kg | 0 | 0 | 13 | 13
  ≥ 35 - < 50 kg | 3 | 0 | 4 | 7
  ≥ 50 - < 70 kg | 10 | 0 | 4 | 14
  ≥ 70 kg | 0 | 8 | 0 | 8
Duration of Plaque Psoriasis [Mean (Standard Deviation); unit: Years] | 7.41 (3.190) | 6.96 (4.057) | 2.75 (2.057) | 4.99 (3.611)
Psoriasis Area Severity Index (PASI) [Mean (Standard Deviation); unit: Units on a scale] — The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
  Units on a scale | 18.78 (11.693) | 15.65 (3.430) | 18.09 (6.144) | 17.84 (7.854)
Baseline Body Mass Index (BMI) category [Count of Participants; unit: Participants]
  Healthy Weight | 7 | 1 | 15 | 23
  Overweight | 2 | 1 | 1 | 4
  Obesity | 4 | 6 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE is an adverse event with a start date on or after the date of the first dose of apremilast and no later than 28 days after the last dose of apremilast. An adverse event is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. A serious AE is any untoward AE that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization or in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or constitutes an important medical event. The investigator assessment of severity/intensity of an event was defined as mild, moderate or severe.
Time Frame: From first dose of apremilast until 28 days after the last dose; up to 29 July 2019; median treatment duration for adolescents apremilast 20 mg and 30 mg was 50.00 and 50.57 weeks respectively and for children was 50.00 weeks.
Population: The safety population consisted of all participants who received at least 1 dose of apremilast
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Adolescents: Apremilast 20 mg | Group 1 Adolescents: Apremilast 30 mg | Group 2 Children: Apremilast 20 mg
Number analyzed (Participants) | 13 | 8 | 21
Participants
  Any TEAE | 13 | 7 | 20
  Any Drug Related TEAE | 11 | 6 | 17
  Any Severe TEAE | 1 | 0 | 1
  Any Serious TEAE | 0 | 0 | 1
  Any Serious Drug-Related TEAE | 0 | 0 | 0
  Any TEAE Leading to Drug Interruption | 1 | 0 | 4
  Any TEAE Leading to Drug Withdrawal | 0 | 0 | 2
  Any TEAE Leading to Death | 0 | 0 | 0

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Apremilast
Description: Maximum observed plasma concentration (Cmax) of apremilast. PK parameters were calculated using non-compartmental methods, plasma concentrations and actual blood sampling times from the intensive sampling schedule.
Time Frame: For adolescents, a pre-dose sample prior to morning dose and on Day 14 as well as at hours 1, 2, 3, 5, 8 and 12 post dose; for the children, samples were collected 2 hours at predose (prior to morning dose) and at 2, 5 and 12 hours post morning dose.
Population: The PK population included all enrolled participants who received one dose of apremilast and had evaluable PK data. PK data was considered evaluable if there were measurable drug levels of apremilast in plasma from at least 3 time points that extended over a minimal 5-hour period within 12 hours post a dose, eg, predose, 2 and 8 hours post a dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group 1 Adolescents: Apremilast 20 mg | Group 1 Adolescents: Apremilast 30 mg | Group 2 Children: Apremilast 20 mg
Number analyzed (Participants) | 12 | 8 | 18
ng/mL | 274.272 (34.3) | 410.929 (39.7) | 348.146 (47.4)

3. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Apremilast
Description: Time to maximum observed plasma concentration obtained directly from the observed concentration versus time data. PK parameters were calculated using non-compartmental methods, plasma concentrations and actual blood sampling times from the intensive sampling schedule.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1 Adolescents: Apremilast 20 mg | Group 1 Adolescents: Apremilast 30 mg | Group 2 Children: Apremilast 20 mg
Number analyzed (Participants) | 12 | 8 | 18
hours | 2.467 [1.00 to 3.00] | 3.000 [1.00 to 5.00] | 2.000 [1.90 to 5.00]

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 12 Hours Post Dose of Apremilast (AUC0-12)
Description: Area under the plasma concentration-time curve from time zero to the 12 hours post dose was calculated using non-compartmental methods, plasma concentrations and actual blood sampling times from the intensive sampling schedule.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 1 Adolescents: Apremilast 20 mg | Group 1 Adolescents: Apremilast 30 mg | Group 2 Children: Apremilast 20 mg
Number analyzed (Participants) | 12 | 8 | 17
ng*h/mL | 1799.717 (36.0) | 2901.795 (41.2) | 2544.874 (40.8)

5. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration of Apremilast (AUC0-t)
Description: Area under the plasma concentration-time curve from time zero to the last quantifiable time point and was calculated using non-compartmental methods, plasma concentrations and actual blood sampling times from the intensive sampling schedule.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 1 Adolescents: Apremilast 20 mg | Group 1 Adolescents: Apremilast 30 mg | Group 2 Children: Apremilast 20 mg
Number analyzed (Participants) | 12 | 8 | 18
ng*h/mL | 1794.815 (35.9) | 2900.472 (41.4) | 2367.641 (50.2)

6. Primary Outcome: Apparent Total Plasma Clearance When Dosed Orally (CL/F) for Apremilast
Description: Apparent total plasma clearance (CL/F) of apremilast was calculated using non-compartmental methods, plasma concentrations and actual blood sampling times from the intensive sampling schedule.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Group 1 Adolescents: Apremilast 20 mg | Group 1 Adolescents: Apremilast 30 mg | Group 2 Children: Apremilast 20 mg
Number analyzed (Participants) | 12 | 8 | 17
Liters/hour | 11.113 (36.0) | 10.338 (41.2) | 7.859 (40.8)

7. Primary Outcome: Apparent Total Volume of Distribution When Dosed Orally, Based on Study-State (Vss/F) or in the Terminal Phase (Vz/F)
Description: Apparent total volume of distribution when dosed orally, based on study-state (Vss/F) or in the terminal phase (Vz/F). Pharmacokinetic parameters were calculated using non-compartmental methods, plasma concentrations and actual blood sampling times from the intensive sampling schedule.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Group 1 Adolescents: Apremilast 20 mg | Group 1 Adolescents: Apremilast 30 mg | Group 2 Children: Apremilast 20 mg
Number analyzed (Participants) | 12 | 8 | 17
Liters | 86.870 (56.1) | 101.049 (31.6) | 55.126 (51.2)

8. Secondary Outcome: Taste and Acceptability of Apremilast Tablets Using the Faces Likert Scale
Description: Taste and acceptability of the apremilast tablet was assessed using a faces Likert Scale on Day 1, initial dosing. The scale consists of options from 1 (dislike very much, illustrated by a frowning face) to 5 (like very much, illustrated by a smiling face).
Time Frame: Day 1
Population: The Safety Population consisted of all participants who received at least 1 dose of apremilast.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Adolescents: Apremilast 20 mg | Group 1 Adolescents: Apremilast 30 mg | Group 2 Children: Apremilast 20 mg
Number analyzed (Participants) | 13 | 8 | 21
Participants
  1 (Dislike Very Much) | 0 | 0 | 3
  2 (Dislike a Little) | 1 | 0 | 1
  3 (Not Sure) | 5 | 4 | 3
  4 (Like a Little) | 1 | 1 | 4
  5 (Like Very Much) | 6 | 3 | 10

9. Primary Outcome: Terminal Phase Elimination Half-Life
Description: Terminal-phase elimination half-life (t ½). PK parameters were calculated using non-compartmental methods, plasma concentrations and actual blood sampling times from the intensive sampling schedule.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group 1 Adolescents: Apremilast 20 mg | Group 1 Adolescents: Apremilast 30 mg | Group 2 Children: Apremilast 20 mg
Number analyzed (Participants) | 12 | 8 | 17
hours | 5.418 (43.1) | 6.775 (50.3) | 4.862 (30.2)

ADVERSE EVENTS:
Time Frame: From first dose of apremilast until 28 days after the last dose; up to 198 weeks; median treatment duration for adolescents apremilast 20 mg and 30 mg was 50.00 and 50.57 weeks respectively and for children was 50.00 weeks.
Arm/Group | Group 1 Adolescents: Apremilast 20 mg | Group 1 Adolescents: Apremilast 30 mg | Group 2 Children: Apremilast 20 mg
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/8 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/8 | 1/21
Other Adverse Events (participants affected / at risk) | 13/13 | 7/8 | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 Adolescents: Apremilast 20 mg (N=13) | Group 1 Adolescents: Apremilast 30 mg (N=8) | Group 2 Children: Apremilast 20 mg (N=21)
Syncope (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 Adolescents: Apremilast 20 mg (N=13) | Group 1 Adolescents: Apremilast 30 mg (N=8) | Group 2 Children: Apremilast 20 mg (N=21)
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 6 | 1 | 11
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 4
Change of bowel habit (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 4 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 4 | 10
Vomiting (Gastrointestinal disorders) | 4 | 1 | 8
Fatigue (General disorders) | 2 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 2
Gastroenteritis (Infections and infestations) | 2 | 1 | 5
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 1
Influenza (Infections and infestations) | 2 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 3 | 7
Pharyngitis streptococcal (Infections and infestations) | 1 | 1 | 0
Tonsillitis streptococcal (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 2 | 0
Viral infection (Infections and infestations) | 1 | 1 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 1 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 3
Monocyte count increased (Investigations) | 0 | 0 | 2
Protein urine present (Investigations) | 1 | 0 | 2
Weight decreased (Investigations) | 2 | 0 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 7 | 1 | 11
Syncope (Nervous system disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 1
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0 | 1
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (2):
  • Study Protocol (2016-04-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT02576678/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT02576678/SAP_001.pdf